CLINICAL TRIAL: NCT01843881
Title: The Contribution of Incretin Hormones to Post-prandial Glucose Metabolism After Roux-en-Y Gastric Bypass
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Adrian Vella (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor-Investigator, Adrian Vella, Consultant, Endocrinology, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 11-007667; R01DK082396 (NIH); UL1RR024150 (NIH)
Record Dates: First submitted 2013-04-26; First posted 2013-05-01 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Gastric Bypass; bariatric surgery; carbohydrate metabolism
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — exendin (9-39)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exendin 9, 39 (Experimental): Exendin 9, 39 will be infused at 300pmol/kg/min in either first intervention period or second intervention period.
  Interventions: Drug: Exendin 9, 39
- Placebo (Placebo Comparator): A saline infusion will be administered in either first intervention period or second intervention period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Exendin 9, 39 — Exendin 9,39 is a competitive antagonist of endogenous GLP-1.
  Arms: Exendin 9, 39
Drug: Placebo — A saline infusion will be given to match the study drug infusion.
  Arms: Placebo

SUMMARY:
The study is being undertaken to understand how the Roux-en-Y Gastric Bypass procedure can affect insulin secretion after meals. The hypothesis of this study is the Disposition Index is decreased in subjects who had previously undergone Roux-en-Y Gastric Bypass by glucagon-like peptide-1 (GLP-1) receptor blockade.

ELIGIBILITY:
Inclusion Criteria Roux-en-Y Gastric Bypass (RYGB)Subjects:

* Subjects who have undergone RYGB

Inclusion Criteria Healthy Subjects:

* Must match RYGB subjects in age, weight, and gender
* Subjects will be without active systemic illness

Exclusion Criteria all Subjects:

* Subjects <20 years old and >70 years old
* For Female Subjects: positive pregnancy text at the time of enrollment or study
* Subjects with functional or organic bowel symptoms.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-03; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in Total Disposition Index from Study 1 (Exendin 9,39) to Study 2 (saline) | Day 1, Day 2 (approximately 2 weeks after day 1)
  The total disposition index equals the product of insulin secretion and insulin sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Vella, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States